CLINICAL TRIAL: NCT06505135
Title: Stem Cell Treatment for Regeneration of the Rotator Cuff (Lipo-Cuff Study)
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHS-Ort-1-2004
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Rotator Cuff Tears; Rotator Cuff Injuries; Rotator Cuff Tear Arthropathy
Keywords: Stem cells
MeSH Terms: conditions — Rotator Cuff Injuries; Rotator Cuff Tear Arthropathy | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The study is designed as a prospective, randomized interventional trial to evaluate the effectoutcome of the treatment of rotator cuff tear with combined standard surgical attachment (standard care) of the supraspinatus tendon and supplementary injection of micro-fragmented tissue into the supraspinatus muscle (cell treatment group) compared to standard care only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Active Comparator): ROTATOR CUFF SURGERY Rotator cuff tendon suture is carried out at Hospital Sønderjylland according to inclusion criteria. Standard treatment also includes intravenous injection preoperatively of 2 g of Cloxacillin In case of allergy 1.5 g of Cefuroxim is chosen. Tendon suture is performed arthroscopically under regional anaesthetic blockage and light sedation with standard double row technique using suture anchors.
  Interventions: Other: Standard care
- Stem-cell treatment (Experimental): HARVEST OF ADIPOSE TISSUE Harvest of adipose tissue from abdominal subcutis and the cell preparation will be performed in the approved lipoplasty system.This lipoaspirate will be processed in the dedicated adipose tissue-processing device. Cell clusters collected at the top of the adipose tissue-processing device undergo a second size reduction by being passed through a size reduction filter. The final product (approximately 60-100 mL) is then concentrated and collected into a 10-mL syringe for subsequent use.
  HARVEST OF MUSCLE BIOPSY FROM THE SUPRASPINATUS MUSCLE A biopsy of 0.1-0.2 g muscle is obtained from the supraspinatus muscle to estimate preoperative muscle fiber atrophy, intracellular lipid accumulation, mitochondrial dysfunction, inflammation and reduced regenerative capacity. The muscle biopsy specimens will be taken near the muscular tendinous junction during routine exposure or arthroscopy of the glenohumeral region.
  Interventions: Biological: Stem-cell treatment

INTERVENTIONS:
Biological: Stem-cell treatment — In the cell treatment group of patients, injection of the cell suspension will be performed at the end of the surgical procedure. Fluid is carefully aspirated via the anterior outflow cannula, and autologous micro-fragmented adipose tissue is injected in dry arthroscopy conditions from the lateral portal while maintaining a subacromial view from the posterior portal.
  10 mL of the stem cells suspension will be injected into the supraspinatus muscle at four predefined sites at the musculo-tendinous junction of the supraspinatus muscle. For each injection site, 1.5 mL of the suspension will be injected using an 18-gauge syringe.
  Arms: Stem-cell treatment
Other: Standard care — Standard treatment also includes intravenous injection preoperatively of 2 g of Cloxacillin In case of allergy 1.5 g of Cefuroxim is chosen. Tendon suture is performed arthroscopically under regional anaesthetic blockage and light sedation with standard double row technique using suture anchors
  Arms: Standard Care

SUMMARY:
Treatment of rotator cuff tears with micro-fragmented adipose tissue is a minimal-invasive procedure with the potential to shorten and ease recovery, accelerate return to daily activity and work of thus with a potential capacity to improve the functional result compared to conventional surgery alone. The study will provide evidence whether the addition of micro-fragmented adipose tissue therapy can augment conventional rotator cuff tear treatment. The study will also reveal whether this treatment can be feasible for standard care of patients with rotator cuff tear as it will be simple to standardize. Moreover, besides providing a novel treatment for patients with rotator cuff tears, the project will based on data from muscle biopsies and scanning modalities, generate new knowledge, preparing for precision regenerative medicine in shoulder disease.

DETAILED DESCRIPTION:
Damage to the tendons that stabilize the shoulder, particularly the supraspinatus tendon tear, has been recognized as the key lesion in rotator cuff tears. However, the lack of full functional recovery after surgical tendon reconstruction suggests that additional changes in the tissue are obstacles to rehabilitation. Recent studies demonstrate pathological changes in the supraspinatus muscle in animal models as a consequence of tendon tear. The muscle pathology includes muscle fibre atrophy, intracellular lipid accumulation, mitochondrial dysfunction, fibril disorganization, and reduced regenerative capacity. Moreover, fibrosis, accumulation of adipocytes, and inflammation develop in these muscles. Muscle strength is decreased by 30% several months after rotator cuff tear repair. Thus, the muscle becomes weaker and stiffer despite repair, suggesting that treatment of rotator cuff tear should include managing cuff muscle dysfunction.

Adipose derived cell therapy Muscle regeneration occurs in a specific environment to which several cell types contribute. The resident stem cell in skeletal muscle is the satellite cell. When skeletal muscle is damaged, the satellite cells are activated and start to proliferate to muscle repairing myoblast. Additional cell types support the regeneration by modulating the myoblast response, inflammation and vascularization. Skeletal muscle harbours a mesenchymal cell, the Fibro-Adipogenic Progenitor (FAP) cell. We have shown that FAPs respond to muscle damage, and is part of the muscle stem cell niche with supportive functions in muscle regeneration. This makes the use of FAPs or mesenchymal cells with a similar function derived from fat an interesting approach for muscle repair.

Implantation of various preparations of cell material that contain Mesenchymal Stromal Cells (MSC) have been used as therapy in a wide range of disorders including lesions in cardiac muscle. The most common sources of cells have been the bone marrow and adipose tissue, and the preparations have ranged from crude isolates of mononuclear cells, e.g. total stromal cells to more homogenous cultured cell isolates, that mainly contain MSC. Although these mesenchymal cells are able to differentiate into tissues such as bone and fat18, their major implication in tissue repair appears to be a capacity to support the regenerative milieu. Their known capacities include stimulation of tissue-specific cells like the myogenic cells, induction of vessel growth, and regulation of inflammation and apoptosis. Cells extracted from adipose tissue cells have shown a regenerative effect without major adverse effects when used as therapy in a range of tissue. Compared to skeletal muscle it is easier and less traumatic to obtain regenerative cells in a sufficient quantum from adipose tissue.

Production of cell preparations exclusively consisting of MSC requires isolation procedures and culturing for weeks, all of which has to be performed in certified laboratories. In case of homolog transplantation, the patient will have to have tissue harvested weeks before the operation. However, cell preparations enriched with MSC can be manufactured with simple, physical treatment of aspirated adipose tissue in a closed system. This can take place in the operation theatre within an hour. This means, that the preparation can be performed the same day as the implantation shall take place, in connection with the main operation.

The adipose tissue will be processed with cutting, grinding, and filtering - not to be considered as substantial manipulation. Likewise, the expected functions of the implanted, active cells in muscle are also found in adipose tissue, which is why the material probably not should be considered as engineered.

The material is derived from adipose tissue and will be used in skeletal muscle, and the use can in this respect be considered non-homologous. However, as the expected major functions in skeletal muscle are the same as in adipose tissue, the function may be accepted as homologous.

Therefore this trial treats patients in a one-day procedure. The adipose tissue will be harvested and processed as an initial procedure during surgery. At the end of the tendon suture procedure, the MSC enriched fragmented tissue will be injected into the supraspinatus muscle.

ELIGIBILITY:
Inclusion Criteria

* Clinical signs and symptoms compatible with a traumatic RCT
* MR verified supraspinatus tear
* Reparable lesion with tendon retraction < 2 cm.
* Fatty infiltration level 0-2 (out of 5) according to Fuchs et al. and based on Goutalliers classification
* No history of inflammatory disease
* ASA score < 3 (patients in good health)
* Signed consent to the study (including use of relevant data from the patient's electronic health records)

Exclusion Criteria

* No MRI of the shoulder
* Former surgery in the affected shoulder
* Signs of infection
* Immunosuppression (due to clinical condition or medical therapy)
* History of inflammatory disease
* Malignancy within 5 years
* Previous radiotherapy to the shoulder
* BMI under 18
* BMI above 35
* Coagulopathy
* Non-Danish speaking patients

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Patient reported outcome of Oxford shoulder score | From inclusion and until 12 months after operation
  A difference in 8 points from the oxford shoulder score questionnaire. The Oxford Shoulder Score comprises twelve items: four assessing the degree of pain and eight evaluating function. Each item is rated on a 5-point Likert scale, where 0 indicates the worst outcome, and 4 indicates the best. The scores from these 12 items are summed to produce a total score ranging from 0 to 48

SECONDARY OUTCOMES:
Clinical healing of the shoulder | 12 months post surgery
  Defined as pain-free movement above shoulder level
Radiological healing | baseline, 6 and 12 months post-surgery
  Defined as closure of the gap between the tendon and the greater tuberosity that serves as the attachment for rotator cuff muscles assessed by MRI .
Functioning of the supraspinatus muscle with improved muscle strain | baseline, 3, 6 and 12 months post-surgery
  Recorded be speckle tracking ultrasonography.
Oxford shoulder score | baseline, 3, 6 and 12 months post-surgery
  Difference in points measured by the oxford shoulder score
Quality of life (EQ5D) | baseline, 3, 6 and 12 months post-surgery
  Difference in points measured by EQ5D questionnaire. The EuroQol-5 Dimension (EQ-5D-5L): Improvements from the baseline in the EQ-5D-5L include self-rated health by a visual analog scale (VAS) measured by 3, 6, and 12 months. The EQ5D measures the quality of life on a 5-point Likert scale based on mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, ranging from "no problems" to "extreme problems" . A key feature of the EQ-5D is the availability of "value sets" that weight the health states reported by patients into utility indexes according to the preferences of a country. For the Danish population, these values range from -0.757 to 1.0, where 1.0 corresponds to absolute health, 0 corresponds to death, and negative values correspond to a health status considered worse than death. The VAS scale is numbered from 0 to 100. 100 means the best health you can imagine. 0 means the worst health you can imagine.

CONTACTS AND LOCATIONS:
Overall Officials: Lars H. Frick, Prof., Principal Investigator — University of Hospital of Southern Denmark - Aabenraa
Locations (1):
- Orthopaedic Research Unit, Department of Orthopaedics, Hospital Sønderjylland, Region of Southern Denmark., Sønderborg, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cartuliares MB, Hejbol EK, Schroder HD, Pedersen AK, Frich LH. Stem cell treatment for regeneration of the rotator cuff: study protocol for a prospective single-center randomized controlled trial (Lipo-cuff). Trials. 2024 Oct 19;25(1):696. doi: 10.1186/s13063-024-08557-0. PMID 39427182